CLINICAL TRIAL: NCT01164657
Title: A Swedish Randomized Controlled Trial of Birth on a Birthing Seat
Brief Title: A Swedish Trial of Birth on a Birthing Seat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsingborgs Hospital (Other)
Collaborators: Stig and Ragna Gorthons foundation (Unknown)
Responsible Party: Li Thies-Lagergren, Reg. Midwife, Mmid, Helsingborgs Hospital, Sweden
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2005/214
Record Dates: First submitted 2009-03-04; First posted 2010-07-19 (Estimated); Last update posted 2010-07-19 (Estimated); Status verified 2009-08

CONDITIONS: Parturition
Keywords: upright position; birth position; childbirth; instrumental deliveries; primiparous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- study group (Experimental): Randomized to give birth on a birthing seat
  Interventions: Device: "BirthRite"
- control group (No Intervention): Randomized to birth in any other position except the birthing seat
  Interventions: Device: "BirthRite"

INTERVENTIONS:
Device: "BirthRite" — Randomization takes place on admission to delivery unit, study group participants seated on the birthing seat when cervix is fully dilated.
  Other Names: "BirthRite" birthing seat

SUMMARY:
Background:

The World Health Organization (WHO) advises against recumbent or supine position for longer periods during labour and birth and states that caregivers should encourage and support the woman to take the position she finds most comfortable. It has been suggested that upright positions may improve childbirth outcomes and reduce the risk for instrumental delivery.

Objective:

The primary objective was to test the hypothesis that birthing on the "BirthRite" ® seat will result in a reduction in the number of primiparous women delivered instrumentally.

Method:

A power calculation showed (α = 0.05 β = 0.2) a requirement of 460 participants in each of the two arms of the trial in order to test for a 40% reduction (from 15% to 9%) of instrumental deliveries in primiparous women at a maternity unit in southern Sweden. It was decided to subject the study to a feasibility test by conducting a pilot-study in which 68 women were randomised to give birth on the birthing seat or to give birth in any other position but on the "BirthRite" ® seat. Randomization to birth on the birthing seat or in any other position took place when the participant's cervix was fully dilated. The primary outcome measurement was the number of instrumental deliveries. Secondary outcome measurements included oxytocin augmentation, perineal trauma, and blood loss administration of oxytocin for augmentation of labour, length of the second stage of labour, perineal trauma, perineal oedema, maternal blood loss and haemoglobin, apgar scores, cord pH and transfers to the Neonatal Intensive Care Unit(NICU).

ELIGIBILITY:
Inclusion Criteria:

* The pilot study included primiparous women who understood the Swedish language sufficiently well to receive information and give informed consent or refusal for participation.
* Pregnancy must have been normal, with a singleton fetus in cephalic presentation and the onset of labour occurring between gestation weeks 37 + 0 and 41 + 6.
* Women having diet treated pregnancy diabetes were also included.
* Obstetric primiparous women with former caesarean section were included as well as those induced because of premature rupture of membranes (PROM).

Exclusion Criteria:

* Multiparous women were excluded from the pilot study.
* Primiparous women were excluded in cases of birth before week 36 + 6, breech presentation, maternal BMI over 30, multiple pregnancy or infectious disease.
* Primiparous women with pre-eclampsia or other conditions that require medical care were not eligible for the pilot study.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2005-11; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Number of women delivered instrumentally | Information collected for each individual 2 hours after delivery. Material collected and analysed at completion of the study (May, 2006)

SECONDARY OUTCOMES:
Administration of oxytocin for augmentation of labor | Information collected for each individual, 2 hours after delivery. Material collected and summarised at completion of study (May, 2006).

CONTACTS AND LOCATIONS:
Overall Officials: Claes Lindoff, PhD, MD, Study Director — Helsingborgs Hospital; Linda J Kvist, PhD, RM, Study Chair — Helsingborgs Hospital
Locations (1):
- Helsingborgs Hospital, Helsingborg, Skåne County, Sweden